CLINICAL TRIAL: NCT02422810
Title: Characterization of a Novel High-Shear Thrombosis Assay in Normal and Aspirin-treated Patients
Brief Title: High-Shear Microfluidic Thrombosis Assay
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sharon Horesh Bergquist, Assistant Professor, Emory University
Other Study IDs: IRB00075811
Record Dates: First submitted 2015-04-17; First posted 2015-04-21 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Coagulation Defects, Other and Unspecified
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No aspirin: Subjects who have not taken aspirin or other blood thinners in the previous 10 days
- Aspirin Daily: Subjects who have taken aspirin daily for the previous 10 or more days
- New to aspirin: Subjects newly started on aspirin during their visit

SUMMARY:
The purpose of this study is to characterize a new test to assess the rate and time it takes to form a blood clot in people who either do or do not take aspirin.

DETAILED DESCRIPTION:
It is estimated that approximately 25% of people are resistant to aspirin, or do not respond to its effect. These individuals have a four fold higher risk of a heart attack or stroke compared to those who respond to aspirin. Current tests for determining those who are aspirin resistant are not reliable. This study is assessing the effectiveness of a new assay in determining the rate and time it takes for people who are or are not on aspirin in forming a blood clot.

ELIGIBILITY:
Inclusion Criteria for "no aspirin" group:

* have not taken aspirin, other nonsteroidal anti-inflammatory drugs (NSAIDs), or clopidogrel in the previous 10 days
* no history of myocardial infarction, ischemic stroke, or other ischemic event

Inclusion Criteria for "aspirin daily" group:

* have taken aspirin daily over the last 10 days or more
* no history of myocardial infarction, ischemic stroke, or other ischemic event

Inclusion Criteria for "new to aspirin" group:

* have not previously been prescribed aspirin, but have been prescribed aspirin at their present appointment, e.g. a high calcium plaque score on CT
* no history of myocardial infarction, ischemic stroke, or other ischemic event

Exclusion Criteria:

* a known bleeding or thrombotic disorder

Exclusion Criteria for "new to aspirin" group:

* a known bleeding or thrombotic disorder
* have taken aspirin, other NSAIDs, clopidogrel, or an anticoagulant in the previous 10 days

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are healthy Emory Executive Health patients over the age of 45 with no history of myocardial infarction, ischemic stroke, or other ischemic event
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Thrombotic occlusion time | 30 minutes
  A microfluidic assay will be used to assess thrombus formation induced by exposed collagen within a stenosis that induces high shear rates. The amount of time taken to completely occlude an aperture is called the thrombotic occlusion time.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bergquist, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States